CLINICAL TRIAL: NCT04205123
Title: Academic Multicenter Prospective Observational Study of the Factors Responsible for Nephropathy in Patients With Sickle Cell Disease Followed by Belgium and the Nord-Pas -De- Calais Region and Creating a Biobank of Blood and Urine
Brief Title: Biological, Genetic and Environmental Involved in the Complications of Sickle Cell Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2014/251
Record Dates: First submitted 2014-10-08; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; nephropathy
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases | interventions — Hemoglobin, Sickle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sickle cell syndrome: Inclusions of sickle cell patients aged over 17 years followed regularly in the participating centers.
  Interventions: Genetic: sickle cell syndrome

INTERVENTIONS:
Genetic: sickle cell syndrome — Academic Study prospective multicenter observational factors responsible for nephropathy in patients with sickle cell disease followed by Belgium and the Nord-Pas -De- Calais Region and creating a biobank of blood and urine.
  In the population of patients with SCD followed in all participating centres.
  Know the prevalence of nephropathy and the relationship between it with their some of their genotypic mutations and clinical phenotype promoting mutated hemoglobin polymerization.
  Determine the behaviour of dense cells in the basal state and in a hypeosmolaire environment
  Determine the place of the erythrocyte microparticles as a biomarker of sickle cell nephropathy
  Studying genes known as risk factor for proteinuria
  Create a BioBank of samples of sickle cell patients in clinically stable condition for other research purposes.

SUMMARY:
The objective of the study is to refine our knowledge on the physiopathology of the symptoms and the complications for the patients affected by a drepanocytic syndrome.

The establishment of risk factors and indicators of severity will allow to target better the patients requiring an adequate strategy in order to prevent the installation of some complications or to limit their worsening.

DETAILED DESCRIPTION:
Some additional tubes will be taken during the usual control of blood test of the drepanocytic patient. A sample of urine will be also asked. Tubes, after pre-treatment, will be sent to Erasme hospital.

A series ob biological but also genetic parameters, both at asymptomatic patients and those in aigüe phase of the disease, can be measured either immediately or a little time after the prelevement.

In this way, we can study numerous domains linked to the physiopathology of the drepanocytose (hémolyse, vaso-occlusion, rheology, factors modulators of the clinical expression). The surplus of the collection could be used for other researchs. It's in this context that we also wish to constitute a biobank of serum, plasma and urine for these drepanocytic patients by surplus of taken material.

The study is realized within the framework of an academic collaboration between institutions. The bank of takings will be located in the reference center of the pathologies of the Red Blood Cell (laboratory of medical chemistry of the erasme hospital).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with sickle cell syndrome
* Signing an inform consent form after validation on it by the Ethics Committees of the participating centers.

Exclusion Criteria:

* Any pathology concomitant risk of nephropathy
* Severe CVO within the month preceding the sampling
* Transfusions within 3 months prior to sampling
* Pregnant patient or within 3 months post- accouhcement

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will characterize the population of sickle cell patients 17 years and older , followed by Belgium and the Nord-Pas -De- Calais, and in the study through the signing of an inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10-20; Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Albumin | each year
  Nephropathy Prevalence

SECONDARY OUTCOMES:
Erythrocyte Microparticles | each year
  Sickle cell Nephropathy biomarker
Eythrocyte Deformability and Erythrocyte Agregation | each year
  Sickle Cell Nephropathy Biomarker
Hp, ApoL1 and HO-1 gene | first year of inclusion
  Sickle Cell Nephropathy risk factor

OTHER OUTCOMES:
Urine, Plasma and Serum aliquotes in a biobank | Each year
  For additional projects

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme Hospital, Brussels, Belgium